CLINICAL TRIAL: NCT00134030
Title: A Randomized Trial of the European and American Osteosarcoma Study Group to Optimize Treatment Strategies for Resectable Osteosarcoma Based on Histological Response to Pre-operative Chemotherapy
Brief Title: Combination Chemotherapy, PEG-Interferon Alfa-2b, and Surgery in Treating Patients With Osteosarcoma
Acronym: EURAMOS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); University College, London (Other); Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Babasola (Sola) Popoola, Matthew Sydes, Professor of Clinical Trials and Methodology, University College, London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOST0331/ EURAMOS-1; NCI-2009-01066 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ISRCTN67613327 (Registry Identifier: ISRCTN); MRC-BO08 (Other: MRC CTU); MRC-EURAMOS1 (Other: MRC CTU); 06-93 (Other: Children's Oncology Group); CDR0000438714 (Other: TBC); COG-AOST0331 (Other: Children's Oncology Group); EU-20530 (Other: TBC); 2004-000242-20 (EudraCT Number); AOST0331 (Other: Children's Oncology Group); AOST0331 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Results first posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Localized Osteosarcoma; Metastatic Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Doxorubicin; Etoposide; Ifosfamide; Methotrexate; merphos; peginterferon alfa-2b

ARMS (4):
- Maintenance therapy group 1 arm I (Active Comparator): Patients receive doxorubicin IV continuously over 48 hours on days 1-2 in weeks 12, 17, 22, and 26 and cisplatin IV over 4 hours on days 1 and 2 in weeks 12 and 17. Patients also receive high-dose MTX IV over 4 hours on day 1 in weeks 15, 16, 20, 21, 24, 25, 28, and 29.
  Interventions: Drug: Cisplatin; Drug: Doxorubicin Hydrochloride; Drug: Methotrexate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Therapeutic Conventional Surgery
- Maintenance therapy group 1 arm II (Experimental): Patients receive doxorubicin, cisplatin, and high-dose MTX as in arm I. Patients than receive PEG-interferon alfa-2b subcutaneously once daily on day 1 in weeks 30-104.
  Interventions: Drug: Cisplatin; Drug: Doxorubicin Hydrochloride; Drug: Methotrexate; Biological: Peginterferon Alfa-2b; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Therapeutic Conventional Surgery
- Maintenance therapy group 2 arm I (Active Comparator): Patients receive doxorubicin, cisplatin, and high-dose MTX as in group 1 arm I.
  Interventions: Drug: Cisplatin; Drug: Doxorubicin Hydrochloride; Drug: Methotrexate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Therapeutic Conventional Surgery
- Maintenance therapy group 2 arm II (Experimental): Patients receive doxorubicin IV continuously over 48 hours on days 1-2 in weeks 12, 20, 28, and 36 and cisplatin IV over 4 hours on days 1 and 2 in weeks 12 and 28. Patients also receive high-dose MTX IV over 4 hours on day 1 in weeks 15, 19, 23, 27, 31, 35, 39, and 40. Patients receive ifosfamide IV over 4 hours on days 1-5 in weeks 16, 24, and 32 and on days 1-3 in weeks 20 and 36 and etoposide IV over 1 hour on days 1-5 in weeks 16, 24, and 32.
  Interventions: Drug: Cisplatin; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Ifosfamide; Drug: Methotrexate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
  Arms: Maintenance therapy group 2 arm II
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
  Arms: Maintenance therapy group 2 arm II
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Peginterferon Alfa-2b — Given subcutaneously
  Other Names: PEG Interferon Alpha-2b; PEG Intron; PEG-IFN Alfa-2b; PEG-IFN-a 2b; PEG-Interferon Alfa-2b; PEG-Intron; Pegylated Interferon Alpha-2b; Polyethylene Glycol IFN-A2b; Polyethylene Glycol Interferon Alfa-2b; SCH 54031; Sylatron
  Arms: Maintenance therapy group 1 arm II
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Therapeutic Conventional Surgery — Undergo amputation or limb salvage surgery

SUMMARY:
This randomized phase III trial is studying combination chemotherapy followed by surgery and two different combination chemotherapy regimens with or without PEG-interferon alfa-2b to compare how well they work in treating patients with osteosarcoma. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Biological therapies, such as PEG-interferon alfa-2b, may interfere with the growth of tumor cells. Giving combination chemotherapy before surgery may shrink the tumor so it can be removed. Giving combination chemotherapy together with PEG-interferon alfa-2b after surgery may kill any remaining tumor cells. It is not yet known whether giving combination therapy together with PEG-interferon alfa-2b is more effective than two different combination chemotherapy regimens alone after surgery in treating osteosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare whether adjuvant maintenance therapy comprising doxorubicin, cisplatin, and high-dose methotrexate (MAP) alone vs MAP combined with ifosfamide and etoposide improves event-free survival of patients with resectable high-grade osteosarcoma who achieve a poor histological response (HR) to neoadjuvant induction therapy comprising MAP.

II. Compare whether adjuvant maintenance therapy comprising MAP alone vs MAP and PEG-interferon alfa-2b improves event-free survival of patients with resectable high-grade osteosarcoma who achieve a good HR to neoadjuvant induction therapy comprising MAP.

SECONDARY OBJECTIVES:

I. Compare overall survival of patients treated with these regimens. II. Compare short- and long-term toxicity of these regimens in these patients. III. Compare quality of life of patients treated with these regimens. IV. Compare event-free survival and overall survival of patients with localized osteosarcoma treated with these regimens.

V. Correlate biological or clinical changes with histological response and outcomes in patients treated with these regimens.

VI. Determine outcomes of patients treated with these regimens.

OUTLINE: This is a randomized, controlled, multicenter study.

INDUCTION THERAPY: (MAP; weeks 1-10) Patients receive doxorubicin IV continuously over 48 hours on days 1-2 and cisplatin IV over 4 hours on days 1 and 2 in weeks 1 and 6. Patients also receive high-dose methotrexate (MTX)* IV over 4 hours on day 1 in weeks 4, 5, 9, and 10. Patients then proceed to surgery.

NOTE: *Patients must receive >= 2 but =< 6 doses of high-dose MTX.

SURGERY: Patients undergo amputation or limb salvage surgery in week 11. Tumor tissue is evaluated for histological response to induction therapy. Patients whose tumor is not amenable to macroscopically complete surgical resection undergo radiotherapy and/or other investigational therapy off study. Patients who undergo macroscopically complete surgical resection of the primary tumor or metastases AND who have no disease progression or unacceptable toxicity proceed to maintenance therapy.

MAINTENANCE THERAPY: Patients are assigned to 1 of 2 groups according to histological response (good [< 10% viable tumor] vs poor [≥ 10% viable tumor]). Patients in each group are stratified according to site of primary tumor and presence of metastases.

GROUP 1: (good histological response) Patient are randomized to 1 of 2 treatment arms within 35 days after surgery.

ARM I: (MAP; weeks 12-29) Patients receive doxorubicin IV continuously over 48 hours on days 1-2 in weeks 12, 17, 22, and 26 and cisplatin IV over 4 hours on days 1 and 2 in weeks 12 and 17. Patients also receive high-dose MTX IV over 4 hours on day 1 in weeks 15, 16, 20, 21, 24, 25, 28, and 29.

ARM II: (MAPifn; weeks 12-104) Patients receive doxorubicin, cisplatin, and high-dose MTX as in arm I. Patients than receive PEG-interferon alfa-2b subcutaneously once daily on day 1 in weeks 30-104.

GROUP 2: (poor histological response) Patients are randomized to 1 of 2 treatment arms within 35 days after surgery.

ARM I: (MAP; weeks 12-29) Patients receive doxorubicin, cisplatin, and high-dose MTX as in group 1 arm I.

ARM II: (MAPIE; weeks 12-40) Patients receive doxorubicin IV continuously over 48 hours on days 1-2 in weeks 12, 20, 28, and 36 and cisplatin IV over 4 hours on days 1 and 2 in weeks 12 and 28. Patients also receive high-dose MTX IV over 4 hours on day 1 in weeks 15, 19, 23, 27, 31, 35, 39, and 40. Patients receive ifosfamide IV over 4 hours on days 1-5 in weeks 16, 24, and 32 and on days 1-3 in weeks 20 and 36 and etoposide IV over 1 hour on days 1-5 in weeks 16, 24, and 32.

In both groups, treatment continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed periodically.

After completion of study treatment, patients are followed every 1½-3 months for 2 years, every 2-4 months for 2 years, every 6 months for 6 years, and then every 6-12 months thereafter. Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade osteosarcoma, including second malignancies

  * Localized or metastatic disease
  * The primary tumor must be located in the limbs or axial skeleton, including any of the following sites*:

    * Long bone of upper limb
    * Short bone of upper limb
    * Long bone of lower limb
    * Short bone of lower limb
    * Vertebral column
    * Ribs, sternum, clavicle, or scapula
    * Pelvic bones, sacrum, or coccyx
* Tumor (primary, metastatic, or both) resectable OR is expected to become resectable after neoadjuvant induction chemotherapy
* Suitable for neoadjuvant chemotherapy
* Performance status - Lansky 50-100% (for patients under 16 years of age)
* Performance status - Karnofsky 50-100%*
* Performance status - WHO or ECOG 0-2*
* Platelet count ≥ 100,000/mm³
* Neutrophil count ≥ 1,500/mm³
* WBC ≥ 3,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal
* Creatinine clearance ≥ 70 mL/min
* Creatinine based on age as follows:

  * No greater than 1.0 mg/dL (for patients 5 to 10 years of age)
  * No greater than 1.2 mg/dL (for patients 11 to 15 years of age)
  * No greater than 1.5 mg/dL (for patients over 15 years of age)
* Ejection fraction ≥ 50% by radionuclide angiogram
* Shortening fraction ≥ 28% by echocardiogram
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity
* No prior chemotherapy for any disease
* Prior radiotherapy for another malignancy allowed
* No prior treatment for osteosarcoma
* No patients with any of the following:

  * Craniofacial osteosarcoma

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1334 (Actual)
Dates: Start 2005-11-14 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neyssa M Marina, Principal Investigator — Children's Oncology Group
Locations (218):
- United States (186):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Harbor-University of California at Los Angeles Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Beaumont Children's Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Cabell-Huntington Hospital, Huntington, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - John Hunter Children's Hospital, Newcastle, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Victoria Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- New Zealand (3):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
  - Wellington Children's Hospital, Wellington
- San Jorge Children's Hospital, San Juan, Puerto Rico
- Switzerland (3):
  - Swiss Pediatric Oncology Group - Bern, Bern
  - Swiss Pediatric Oncology Group - Geneva, Geneva
  - Swiss Pediatric Oncology Group - Lausanne, Lausanne

REFERENCES:
- [Derived] Hazewinkel AD, Lancia C, Anninga J, van de Sande M, Whelan J, Gelderblom H, Fiocco M. Disease progression in osteosarcoma: a multistate model for the EURAMOS-1 (European and American Osteosarcoma Study) randomised clinical trial. BMJ Open. 2022 Mar 4;12(3):e053083. doi: 10.1136/bmjopen-2021-053083. PMID 35246418
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- [Derived] Marina NM, Smeland S, Bielack SS, Bernstein M, Jovic G, Krailo MD, Hook JM, Arndt C, van den Berg H, Brennan B, Brichard B, Brown KLB, Butterfass-Bahloul T, Calaminus G, Daldrup-Link HE, Eriksson M, Gebhardt MC, Gelderblom H, Gerss J, Goldsby R, Goorin A, Gorlick R, Grier HE, Hale JP, Hall KS, Hardes J, Hawkins DS, Helmke K, Hogendoorn PCW, Isakoff MS, Janeway KA, Jurgens H, Kager L, Kuhne T, Lau CC, Leavey PJ, Lessnick SL, Mascarenhas L, Meyers PA, Mottl H, Nathrath M, Papai Z, Randall RL, Reichardt P, Renard M, Safwat AA, Schwartz CL, Stevens MCG, Strauss SJ, Teot L, Werner M, Sydes MR, Whelan JS. Comparison of MAPIE versus MAP in patients with a poor response to preoperative chemotherapy for newly diagnosed high-grade osteosarcoma (EURAMOS-1): an open-label, international, randomised controlled trial. Lancet Oncol. 2016 Oct;17(10):1396-1408. doi: 10.1016/S1470-2045(16)30214-5. Epub 2016 Aug 25. PMID 27569442
- [Derived] Whelan JS, Bielack SS, Marina N, Smeland S, Jovic G, Hook JM, Krailo M, Anninga J, Butterfass-Bahloul T, Bohling T, Calaminus G, Capra M, Deffenbaugh C, Dhooge C, Eriksson M, Flanagan AM, Gelderblom H, Goorin A, Gorlick R, Gosheger G, Grimer RJ, Hall KS, Helmke K, Hogendoorn PC, Jundt G, Kager L, Kuehne T, Lau CC, Letson GD, Meyer J, Meyers PA, Morris C, Mottl H, Nadel H, Nagarajan R, Randall RL, Schomberg P, Schwarz R, Teot LA, Sydes MR, Bernstein M; EURAMOS collaborators. EURAMOS-1, an international randomised study for osteosarcoma: results from pre-randomisation treatment. Ann Oncol. 2015 Feb;26(2):407-14. doi: 10.1093/annonc/mdu526. Epub 2014 Nov 24. PMID 25421877

RESULTS

PARTICIPANT FLOW:
Groups:
- MAP-GR: Patients receive doxorubicin IV continuously over 48 hours on days 1-2 in weeks 12, 17, 22, and 26 and cisplatin IV over 4 hours on days 1 and 2 in weeks 12 and 17. Patients also receive high-dose MTX IV over 4 hours on day 1 in weeks 15, 16, 20, 21, 24, 25, 28, and 29.
  Cisplatin: Given IV
  Doxorubicin Hydrochloride: Given IV
  Methotrexate: Given IV
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Therapeutic Conventional Surgery: Undergo amputation or limb salvage surgery
- MAPifn: Patients receive doxorubicin, cisplatin, and high-dose MTX as in arm I. Patients than receive PEG-interferon alfa-2b subcutaneously once daily on day 1 in weeks 30-104.
  Cisplatin: Given IV
  Doxorubicin Hydrochloride: Given IV
  Methotrexate: Given IV
  Peginterferon Alfa-2b: Given subcutaneously
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Therapeutic Conventional Surgery: Undergo amputation or limb salvage surgery
- MAP-PR: Patients receive doxorubicin, cisplatin, and high-dose MTX as in group 1 arm I.
  Cisplatin: Given IV
  Doxorubicin Hydrochloride: Given IV
  Methotrexate: Given IV
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Therapeutic Conventional Surgery: Undergo amputation or limb salvage surgery
- MAPIE: Patients receive doxorubicin IV continuously over 48 hours on days 1-2 in weeks 12, 20, 28, and 36 and cisplatin IV over 4 hours on days 1 and 2 in weeks 12 and 28. Patients also receive high-dose MTX IV over 4 hours on day 1 in weeks 15, 19, 23, 27, 31, 35, 39, and 40. Patients receive ifosfamide IV over 4 hours on days 1-5 in weeks 16, 24, and 32 and on days 1-3 in weeks 20 and 36 and etoposide IV over 1 hour on days 1-5 in weeks 16, 24, and 32.
  Cisplatin: Given IV
  Doxorubicin Hydrochloride: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Methotrexate: Given IV
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Therapeutic Conventional Surgery: Undergo amputation or limb salvage surgery
Period: Overall Study
Arm/Group | MAP-GR | MAPifn | MAP-PR | MAPIE
Started | 359 | 357 | 310 | 308
Completed | 359 | 357 | 310 | 308
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MAP-GR | MAPifn | MAP-PR | MAPIE | Total
Number analyzed (Participants) | 359 | 357 | 310 | 308 | 1334
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14 [11 to 16] | 14 [12 to 16] | 15 [11 to 18] | 15 [12 to 17] | 14 [12 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 147 | 136 | 117 | 548
  Male | 211 | 210 | 174 | 191 | 786
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 2 | 2 | 0 | 5
  Canada | 20 | 9 | 7 | 11 | 47
  United States | 128 | 134 | 142 | 139 | 543
  Australia | 2 | 3 | 3 | 5 | 13
  Switzerland | 8 | 3 | 7 | 7 | 25
  Austria | 2 | 5 | 5 | 8 | 20
  Belgium | 14 | 14 | 9 | 7 | 44
  Czechia | 3 | 0 | 2 | 1 | 6
  Denmark | 2 | 6 | 2 | 2 | 12
  Finland | 0 | 0 | 1 | 2 | 3
  Germany | 85 | 90 | 60 | 63 | 298
  Hungary | 5 | 6 | 5 | 3 | 19
  Ireland | 0 | 0 | 0 | 1 | 1
  Netherlands | 21 | 18 | 16 | 10 | 65
  Norway | 7 | 10 | 12 | 5 | 34
  Sweden | 14 | 10 | 4 | 5 | 33
  United Kingdom | 47 | 47 | 33 | 39 | 166
Site of tumour [Count of Participants; unit: Participants]
  Femur | 179 | 191 | 154 | 166 | 690
  Tibia | 113 | 102 | 75 | 76 | 366
  Fibula | 14 | 20 | 17 | 13 | 64
  Humerus | 36 | 33 | 39 | 27 | 135
  Radius | 5 | 5 | 4 | 6 | 20
  Ulna | 2 | 0 | 2 | 1 | 5
  Scapula/clavicle | 2 | 1 | 3 | 2 | 8
  Pelvis/sacrum | 5 | 5 | 8 | 11 | 29
  Rib | 3 | 0 | 3 | 3 | 9
  Other | 0 | 0 | 5 | 3 | 8
Location of tumour on the bone [Count of Participants; unit: Participants]
  Proximal | 156 | 150 | 114 | 109 | 529
  Diapysis | 13 | 12 | 11 | 12 | 48
  Distal | 180 | 189 | 166 | 168 | 703
  N/A (not long bone) | 10 | 6 | 19 | 19 | 54
Pathological fracture at diagnosis [Count of Participants; unit: Participants]
  No | 321 | 308 | 276 | 270 | 1175
  Yes | 37 | 49 | 34 | 35 | 155
  Data missing | 1 | 0 | 0 | 3 | 4
Lung metastases [Count of Participants; unit: Participants]
  No/possible | 324 | 321 | 272 | 280 | 1197
  Yes | 35 | 36 | 38 | 28 | 137
Histological classification [Count of Participants; unit: Participants]
  Conventional | 320 | 322 | 288 | 289 | 1219
  Telangiectatic | 25 | 20 | 11 | 6 | 62
  Small cell | 2 | 1 | 3 | 2 | 8
  High-grade surface | 3 | 5 | 5 | 6 | 19
  Other | 4 | 2 | 0 | 1 | 7
  Data missing | 5 | 7 | 3 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: EFS is defined as time from randomisation to the first of: death, detection of local recurrence or metastasis, progression of metastatic disease, or detection of a secondary malignancy.
  EFS will be assessed using the logrank test and expressed using hazard ratios with appropriate confidence intervals. Follow up per participant will be assessed for up to 10 years. The 3 year EFS is provided as a summary.
Time Frame: From date of randomization to date of the event.
Measure: Number (95% Confidence Interval); unit: Percentage EFS
Arm/Group | MAP-GR | MAPifn | MAP-PR | MAPIE
Number analyzed (Participants) | 359 | 357 | 310 | 308
Percentage EFS | 74 [69 to 79] | 77 [72 to 81] | 55 [49 to 60] | 53 [47 to 59]
Statistical Analysis 1: Comparison: MAP-GR vs MAPifn; Test type: Superiority; p = 0.214, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.61 to 1.12]
Statistical Analysis 2: Comparison: MAP-PR vs MAPIE; Test type: Superiority; p = 0.86, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.78 to 1.23]
Statistical Analysis 3: Comparison: MAP-PR vs MAPIE; Secondary RMST analysis performed in poor response group, due to evidence of non-proportional hazards; Test type: Superiority; p = 0.69, Difference in RMST; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-3.3 to 4.9]

2. Secondary Outcome: Percentage of Patients With Overall Survival
Description: Overall survival is time from randomization until death from any cause.
  Will be assessed using the logrank test and expressed using hazard ratios with appropriate confidence intervals. Participants will be assessed for up to 10 years. 5 year overall survival is provided as a summary.
Time Frame: From date of randomization to date of death.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MAP-GR | MAPifn | MAP-PR | MAPIE
Number analyzed (Participants) | 359 | 357 | 310 | 308
Percentage of participants | 84 [80 to 88] | 84 [81 to 88] | 68 [63 to 73] | 68 [63 to 73]
Statistical Analysis 1: Comparison: MAP-GR vs MAPifn; Test type: Superiority; p = 0.804, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.69 to 1.33]
Statistical Analysis 2: Comparison: MAP-PR vs MAPIE; Test type: Superiority; p = 0.674, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.81 to 1.39]

3. Secondary Outcome: Toxicity as Measured by Common Terminology Criteria for Adverse Events (CTCAE) v3.0
Description: Percentages of patients experiencing grade 3 and 4 adverse events. These will be compared using chi-square tests or Fisher's exact tests where appropriate.
Time Frame: Adverse events are assessed for up to 10 years per participant.
Population: Adverse events are only analyzed in participants who started treatment and for whom toxicity data were provided.
Measure: Count of Participants; unit: Participants
Arm/Group | MAP-GR | MAPifn | MAP-PR | MAPIE
Number analyzed (Participants) | 356 | 355 | 301 | 298
Participants | 348 | 340 | 287 | 281

ADVERSE EVENTS:
Time Frame: From randomisation until 30 days after last protocol treatment up to 10 years.
Description: The total number of participants represented in the Serious Adverse Events Table is 1,334 (MAP-GR +MAPifn +MAP-PR+MAPIE). On an intention to treat basis, this includes16 patients (across all arms) who did not start treatment or had no adverse event data available.
Arm/Group | MAP-GR | MAPifn | MAP-PR | MAPIE
Serious Adverse Events (participants affected / at risk) | 49/359 | 76/357 | 36/310 | 43/308
Other Adverse Events (participants affected / at risk) | 0/359 | 0/357 | 0/310 | 0/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAP-GR (N=359) | MAPifn (N=357) | MAP-PR (N=310) | MAPIE (N=308)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 7 (11) | 5 (6) | 3 (4) | 10 (17)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATRIAL THROMBOSIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEAFNESS BILATERAL (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BASEDOW'S DISEASE (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THYROIDITIS (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
ANAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
CHILLS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IMPAIRED HEALING (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFUSION SITE THROMBOSIS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 3 (3) | 2 (2) | 6 (7) | 3 (3)
PYREXIA (General disorders) | 4 (7) | 3 (5) | 2 (2) | 2 (2)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VENOOCCLUSIVE LIVER DISEASE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMOPHAGOCYTIC LYMPHOHISTIOCYTOSIS (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
BACTERIAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CATHETER SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 3 (3) | 6 (7) | 3 (3) | 1 (1)
DEVICE RELATED SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ECTHYMA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEBRILE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
H1N1 INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
IMPLANT SITE CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INCISION SITE ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIC INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 2 (3) | 2 (2) | 1 (1)
PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SCALDED SKIN SYNDROME (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WOUND INFECTION (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
CHEMOTHERAPEUTIC DRUG LEVEL INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
DRUG CLEARANCE DECREASED (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA B VIRUS TEST POSITIVE (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
EWING'S SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL CELL CARCINOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANOSMIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL ARTERY EMBOLISM (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
HEMIPLEGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LEUKOENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
STUPOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEVICE FAILURE (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THROMBOSIS IN DEVICE (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MANIA (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEPHROPATHY TOXIC (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL ARTERY DISSECTION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOCARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OPTIC NEUROPATHY (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFUSION SITE ERYTHEMA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEPTIC ARTHRITIS STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VARICELLA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BONE INFARCTION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CYTOTOXIC OEDEMA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSTONIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MONOPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HYPERSENSITIVITY PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
In the good response patients (randomised to MAP-GR or MAPifn), 128 of 357 MAPifn patients completed the planned protocol treatment. Among poor response patients (randomised to MAP-PR or MAPie), 42% of registered patients were not randomised. Further patients were registered to the trial and joined a treatment cohort for follow-up but declined to join the randomisation or were not eligible. The data for these non-randomised patients are not presented here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-09-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT00134030/Prot_SAP_ICF_000.pdf